



## Master Statistical Analysis Plan Checklist for Investigator Initiated Trials

A Phase II Open Label Study of Everolimus in Combination with Anti-estrogen Therapy in Hormone Receptor-Positive HER2-Negative Advanced Breast Cancer

Sponsor: Sarah Cannon Development Innovations

(Innovations)

Study Drug: Everolimus

SCRI Protocol Number: BRE 212

NCT number: 02291913

Prepared By: Innovations Biostats

Date 06DEC2019

Version 2.0, 06 DEC 2019 

Confidential



REFERENCE SOP: CDS-0102

## Statistical Analysis Plan Checklist for Investigator Initiated Trials History of Changes

This document has undergone the following changes:

| Version Number | Version Date | Description of Changes |
|---|---|---|
| 1.0 | 31MAY2018 | Original document |
| 2.0 | 06DEC2019 | Formatting; textual clarifications with respect to protocol; and TFL output duplicate remediation with renumbering |




| 1.1 Objectives | |
|---|---|
| Primary Objective: | To determine the efficacy of everolimus in combination with anti-estrogen therapy in patients with ER and/or PR-positive, HER2-negative advanced breast cancer demonstrating disease progression on prior hormonal therapy as measured by PFS |
| Secondary Objectives: | To determine the safety and tolerability of everolimus with an anti-estrogen therapy in patients with ER and/or PR-positive, HER2-negative advanced breast cancer |
| Exploratory Objectives: | To evaluate the VeriStrat assay in this HR-positive patient population treated with everolimus in combination with anti-estrogen therapy |
| 1.2 Study Design | |
| Study Type | ⊠ Non-Randomized |
| | ☐ Randomized (Allocation Ratio: ) |
| Details | This is a multi-centered, open-labeled, Phase II study in MBC. The patient population includes locally recurrent or MBC patients with cytologically or histologically confirmed hormone receptor-positive breast cancer who have demonstrated disease progression on prior anti-estrogen therapy or therapies. Eligible patients must have evaluable or measurable disease per RECIST v1.1. |
| | Progression Free Survival (PFS), defined as the time from the first day of study drug administration (Day 1) to disease progression (event) as defined by the RECIST v1.1 criteria, or death (event) on study. Patients who are alive and free from disease progression will be censored at the date of last tumor assessment. Patients who receive non-protocol therapy (subsequent therapy) prior to incurring an event will be censored at the date of last tumor assessment prior to the start of subsequent therapy. Patients who do not have a post-baseline tumor assessment will be censored at the date of first treatment (Day 1). |
| | Overall Survival (OS), defined as the time from the first day of study drug administration (Day 1) or death on study. Patients who are alive will be censored at the date of last known date alive. |
| | Duration of Response (DOR), is defined as the time from the first date of CR or PR to disease progression or death as defined by the RECIST v1.1 criteria. Patients who are alive and free from disease progression will be censored at the date of last tumor assessment. Patients who receive non-protocol therapy (subsequent therapy) prior to incurring an event will be censored at the date of last tumor assessment prior to the start of subsequent therapy. Only those patients who achieved CR or PR will be included in the summaries of DOR. |
| | PFS (efficacy primary endpoint), OS and DOR (efficacy secondary endpoints) estimates will be generated using Kaplan-Meier methods, both for all patients enrolled and those patients receiving the MTD. Four month and six month PFS estimates with 95% confidence intervals (CIs), and median PFS and OS with 95% CIs, will be calculated. |
| | Best overall response will be tabulated: CR, PR, SD, PD and not evaluable (NE). |
| | Overall Response Rate (ORR) is defined as the proportion of patients with observed complete response (CR) or partial response (PR) according to the RECIST v1.1 criteria. |
| | Clinical Benefit Rate (CBR) is defined as the proportion of patients with CR, PR or SD x 6 months according to the RECIST v1.1 criteria. |
| | For ORR and CBR, patients without a post-baseline tumor assessment will be classed as not evaluable (NE) and considered as non-responder. |






| | For ORR and CBR, the estimates and the associated 95% CI (based on both asymptotic normal approximation and exact binomial methods) will be calculated. |
|---|---|
| 1.3.2 Randomization | |
| Randomization Type: | ☐ Open-Label ☐ Single Blind ☐ Double-Blind |
| 1.4 Timing of Analysis | |
| Planned Interim Analysis | <ul> <li>□ Cohort Review / Dose Escalation</li> <li>☑ Safety Review</li> <li>□ Interim Efficacy/Safety Analysis</li> <li>□ Independent DMC/DSMB</li> <li>□ Annual Report / Investigator Brochure (IB)</li> </ul> |
| | ☐ Abstract / Scientific Presentation (Oral/Poster) |
| Final Analysis | The final analysis will occur when 42 patients have discontinued treatment, progressed, died or are still on treatment but have at least 12 months of follow-up (time from first treatment until last tumor assessment). |
| 1.5 Responsibilities | |
| Trial Statistician: | Prepare SAP check list and TFL shells Review deliverables produced by Statistical Programmer |
| PK Statistician: | N/A |
| Independent Statistician: | N/A |
| 1.6 Analysis Software | |
| Main statistical analysis: | SAS Version 9.3 or above |
| Other analysis software: | N/A |
| 1.7 Coding | |
| <ul><li>☑ Adverse Events</li><li>☐ Medical History</li></ul> | <ul> <li>✓ MedDRA:</li></ul> |
| <ul><li>☐ Concomitant Medication</li><li>☐ Prior Therapy</li><li>☐ Subsequent/Further Therapy</li></ul> | ☐ WHO-Drug: ☐ Version ☐ Most current release and update coding with new major releases |






| 2 Analysis Population | |
|---|---|
| Intent-To-Treat (ITT) Population definition: | <ul> <li>☐ All patients who have started treatment in the study</li> <li>☐ All patients who have been randomized in the study, regardless of whether they have received any treatment or not</li> <li>☐ All patients who have been randomized and have started treatment in the study</li> <li>☐ Other definition, specify:</li> </ul> |
| Per Protocol (PP) Population to be used in analysis: | ☐ Yes ☐ No If yes, please specify the criteria for exclusion from the PP population: |
| Safety (SAF) Population definition | <ul> <li>☐ All patients who have started treatment in the study. Patients will be analyzed according to the actual treatment they have received.</li> <li>☑ Other definition, specify: All patients who have received any dose of study treatment.</li> </ul> |
| Other Analysis Population definition: | Efficacy Evaluable (EE): All patients who receive at least 1 cycle of study treatment and have at least one post-baseline assessment. (Patients who discontinue treatment during Cycle 1 will not be replaced in the study.) |
| 3 Baseline Value Definitions | |
| | Last value prior to first date of study treatment |
| 4 Efficacy | |
| 4 Efficacy Response Criteria Used: | □ RECIST 1.0 □ RECIST 1.1 □ Cheson 2007 □ Modified RECIST – specify: □ Other criteria, Specify: |






| Efficacy Endpoints: | | | | | |
|---|---|---|---|---|---|
| Zindady Zindpolinto. | | Endpoint | Primary Analysis<br>Population | Other Ana<br>Population | |
| | Primary | PFS | Efficacy Evaluable | Safety | |
| | Secondary | OS, DOR,ORR, CBR | Efficacy Evaluable | Safety | |
| Definition of Terms: | | | | | |
| ⊠ Response | ☐ Complete F | Response + Partial Resp | onse as best observed | response | |
| | ☐ Complete F | Response + Partial Resp<br>ria, specify: | onse, confirmed with | weeks | apart. |
| ☑ Clinical Benefit | Complete F | Response + Partial Resp | onse + Stable Disease | as best obse | erved |
| | | Response + Partial Resp<br>Disease (at least wee | onse (confirmed with<br>eks from start of treatm | weeks apa<br>ent) | art) |
| | <ul><li>☑ Other criteria, specify: (Complete response (CR) + Partial response (PR)</li><li>+ Stable disease (SD) x 6 months)</li></ul> | | | | |
| □ Progression | Disease progression (event) as defined by the RECIST v1.1 or death on study; non-protocol therapy (subsequent therapy) prior to incurring an event will be censored at the date of last tumor assessment prior to the start of subsequent therapy | | | | |
| Subsequent Therapy | Non-protocol therapy prior to incurring an event | | | | |
| ☐ Treatment Failure | N/A | | | | |
| Definition of Endpoints: | Start Date: | Date of Randomization | ☑ Date of First T | reatment | |
| | , , | ecify for all pertinent end | points): | | |
| | Overall Surviva | l: Event = Death | | | 1 |
| | <u> </u> | Situation | Date of Event of | or Censoring | Outcome |
| | | on-study or follow-up | Date of death | | Event |
| | Alive, as of end of study or follow-up Date last known alive Censored | | | | |
| | Status unknown, as of end of study Date last known alive Censored | | | | |
| | Progression-Free Survival: Event = Progression or Death | | | | |
| | | Situation | Date of Event o | | Outcome |
| | No baseline as | | Date of first trea | | Censored |
| | | ed between scheduled visit<br>nd received no subsequent | * | | Event |
| | PD documented between scheduled visits, did not die, but received subsequent therapy prior to incurring progression event Subsequent therapy | | | | |




## BRE 212 Statistical Analysis Plan Checklist

| Death while on-study without previous PD, and received no subsequent therapy | Date of death | Event |
|---|---|---|
| Death while on-study and had previous PD, and received no subsequent therapy | First date of evaluated overall response = PD | Event |
| Death while on-study without previous PD,<br>but received subsequent therapy prior to<br>death event | Date of last evaluable tumor assessment prior to start of subsequent therapy | Censored |
| Death while on-study and had previous PD,<br>but received subsequent therapy prior to PD<br>event | Date of last evaluable tumor assessment prior to start of subsequent therapy | Censored |
| No progression, no death | Date of last evaluable tumor assessment | Censored |
| Treatment discontinuation for adverse event or other non-event reason | Date of last evaluable tumor assessment | Censored |
| <del>-</del> | rval between treatment arms | |
| p-value, specify statistical test. | | |
| Default: Estimates of medians in each treatment arm | | |
| ☑ Other quartiles or percentages of survival required, specify: PFS: @4 months and 6 months: percentages & 95% confidence intervals | | |
| _ | etween treatment arms, unstr | atified |
| 1 _ ` | | |
| Hazard ratio & 95% confidence interval between treatment arms, stratified (specify stratification factor(s)): | | |
| p-value, specify statistical test: | | |
| Median Follow-up: Estimate of median, 25 <sup>th</sup> and 7 <sup>th</sup> quartiles; Follow-up point estimates: @ 4 months, 6 months, and 12 months: percentages & 95% confidence intervals | | |
| | | n of therapy |
| Data will be summarized by: | | |
| ☐ NCI-CTCAE for CTCAE-gradable parameter | ters, and H/L for non-CTCAE | -Gradable |
| ☐ H/L for all lab parameters | | |
| | Death while on-study and had previous PD, and received no subsequent therapy Death while on-study without previous PD, but received subsequent therapy prior to death event Death while on-study and had previous PD, but received subsequent therapy prior to death event Death while on-study and had previous PD, but received subsequent therapy prior to PD event No progression, no death Treatment discontinuation for adverse event or other non-event reason Default: Estimates of rates in each treatment □ Difference in rates & 95% confidence interest in p-value, specify statistical test: □ Default: Estimates of medians in each treatment in p-value, specify statistical test: □ Hazard ratio & 95% confidence interval be stratification factor(s)): □ p-value, specify statistical test: Median Follow-up: Estimate of median, 25th a Follow-up point estimates: @ 4 months, 6 meconfidence intervals Definition of Treatment-Emergent Adverse Entreatment-emergent AEs are those with an Data will be summarized by: □ NCI-CTCAE for CTCAE-gradable parameter parameter | Death while on-study and had previous PD, and received no subsequent therapy Death while on-study without previous PD, but received subsequent therapy prior to death event Death while on-study without previous PD, but received subsequent therapy prior to death event Death while on-study and had previous PD, but received subsequent therapy prior to PD event Death while on-study and had previous PD, but received subsequent therapy prior to PD event No progression, no death Date of last evaluable tumor assessment prior to start of subsequent therapy No progression, no death Date of last evaluable tumor assessment Treatment discontinuation for adverse event or other non-event reason Default: Estimates of rates in each treatment arm Difference in rates & 95% confidence interval between treatment arms p-value, specify statistical test: Default: Estimates of medians in each treatment arm Mother quartiles or percentages of survival required, specify: PFS: @4 months and 6 months: percentages & 95% confidence interval between treatment arms, unstread p-value, specify statistical test: Hazard ratio & 95% confidence interval between treatment arms, unstread stratification factor(s)): p-value, specify statistical test: Hazard ratio & 95% confidence interval between treatment arms, stratification factor(s)): p-value, specify statistical test: Median Follow-up: Estimate of median, 25th and 7th quartiles; Follow-up point estimates: @ 4 months, 6 months, and 12 months: percent confidence intervals Definition of Treatment-Emergent Adverse Event (TEAE): Treatment-emergent AEs are those with an onset on or after the initiation bata will be summarized by: NCI-CTCAE for CTCAE-gradable parameters, and H/L for non-CTCAE parameter |




## Tier 1 Study – Tables, Figures & Listings

| Standard 7 | Standard TFLs | | |
|---|---|---|---|
| Table No | Description | Variables/Analyses To Be Included | Population |
| Table 1 | Patient Disposition | <ul> <li>Number of patients screened</li> <li>Number of patients enrolled</li> <li>Number of patients treated</li> <li>Reason for treatment discontinuation</li> <li>Reason for study discontinuation</li> <li>Other, specify:</li> </ul> | Enrolled Patients |
| Table 2 | Demographic Characteristics | <ul> <li>Age: N, Mean, SD, Median, Min, Max</li> <li>Age Group: &lt;65, &gt;=65</li> <li>Sex</li> <li>Race</li> <li>Ethnicity</li> <li>ECOG</li> <li>Other, specify:</li> </ul> | Enrolled Patients |
| Table 3 | Disease History - General | <ul> <li>☐ Histology</li> <li>☐ Disease staging at initial diagnosis</li> <li>☐ Time from initial diagnosis to first dose</li> <li>☐ Number of patients with metastatic disease</li> <li>☐ Sites of metastases</li> <li>☐ Other, specify: Histology Grade</li> </ul> | Enrolled Patients |
| Table 4 | Prior Hormonal Therapy | Time [months] from last hormonal therapy to first date of study treatment: N, Mean, SD, Median, Min, Max | Safety |
| Table 5 | Treatment and Dose Modifications | Duration on Treatment (weeks), N, Mean, SD, Median, Min, Max Dose Reduction (n, %) None Patients with 1 Patients with 2 Patients with >= 3 Dose Interruption (n, %) None Patients with 1 Patients with 2 Patients with 2 Patients with >= 3 | Safety |
| Table 6 | Measurable Lesions | Measurable Lesions (n, %) Non-Measurable Lesions (n, %) Evaluable Bone Only Disease (n, %) | Enrolled Patients |
| Table 7 | Best Overall Response | Best overall response (n, %): Complete response (CR), Partial response (PR), Stable disease (SD), NonCR/NonPD, Progressive disease (PD), Not evaluable (NE), Not applicable (N/A) Missing Objective Response Rate (ORR) (= CR+PR): ORR, 95% Confidence interval Clopper-Pearson | Efficacy Evaluable,<br>Safety |




| Standard TFLs | | | |
|---|---|---|---|
| Table No | Description | Variables/Analyses To Be Included | Population |
| | | Normal Approximation Clinical Benefit Rate (CBR) (=CR+PR+SD>=4months): CBR, 95% Confidence interval Clopper-Pearson Normal Approximation Clinical Benefit Rate (CBR) (=CR+PR+SD>=6months): CBR, 95% Confidence interval Clopper-Pearson Normal Approximation] | |
| Table 8 | Progression-free Survival<br>(Kaplan-Meier estimates & 95% CI) | Number of patients with events, Number of patients censored, Median Progression-free Survival [months (95% CI)] 25% Percentile Follow-up [months (95% CI)] 75% Percentile Follow-up [months (95% CI)] Progression-free Survival Estimates [probability, (95% CI)]: 4 months, 6 months, 12 months | Efficacy Evaluable,<br>Safety |
| Table 9 | Overall Survival<br>(Kaplan-Meier estimates & 95% CI) | Number of patients with events, Number of patients censored, Median Overall Survival [months (95% CI)] 25% Percentile Follow-up [months (95% CI)] 75% Percentile Follow-up [months (95% CI)] Overall Survival Estimates [probability, (95% CI)]: 4 months, 6 months, 12 months | Efficacy Evaluable,<br>Safety |
| Table 10 | Adverse Event Overview | Any Adverse Event Treatment-related Adverse Event Everolimus-related Adverse Event Anti-Estrogen Therapy-related Adverse Event Serious Adverse Event Treatment-related Serious Adverse Event Serious Adverse Event leading to Death Treatment-related Serious Adverse Event leading to Death Adverse Events leading to Treatment Discontinuation Adverse Events leading to Treatment Interruption Adverse Events leading to Treatment Reduced | Safety |




REFERENCE SOP: CDS-0102

| Standard TFLs | | | |
|---|---|---|---|
| Table No | Description | Variables/Analyses To Be Included | Population |
| Table 11 | Any Treatment-Emergent Adverse Event<br>by System Organ Class and Preferred<br>Term | System organ class, Preferred term, CTCAE grade [all statistics: (n, %)] | Safety |
| Table 12 | Any Treatment Related-Emergent<br>Adverse Event by System Organ Class<br>and Preferred Term | System organ class, Preferred term, CTCAE grade [all statistics: (n, %)] | Safety |
| Table 13 | Any Treatment Related-Emergent<br>Adverse Event by SCRI Grouped<br>Adverse Event Term | SCRI grouped AE term,<br>CTCAE grade<br>[all statistics: (n, %)] | Safety |
| Table 14 | Treatment Serious-Emergent Adverse<br>Event by System Organ Class and<br>Preferred Term | System organ class, Preferred term, CTCAE grade [all statistics: (n, %)] | Safety |
| Table 15 | Treatment Related and Serious-<br>Emergent Adverse Event by System<br>Organ Class and Preferred Term | System organ class, Preferred term,<br>CTCAE grade<br>[all statistics: (n, %)] | Safety |
| Table 16 | Duration of Response (DOR)<br>(Kaplan-Meier estimates & 95% CI) | Number of patients with events, Number of patients censored, Duration of Response: Median [months (95% CI)] | Efficacy Evaluable,<br>Safety |
| | | Duration of Response Estimates<br>[probability, (95% CI)]:<br>4 months, 6 months | |
| Table 17 | Median Follow-up<br>(Kaplan-Meier estimates & 95% CI) | Number of patients with events, Number of patients censored, Median Follow-up [months (95% CI)] 25% Percentile Follow-up [months (95% CI)] 75% Percentile Follow-up [months (95% CI)] | Efficacy Evaluable |
| | | Follow-up Estimates<br>[probability, (95% CI)]:<br>4 months, 6 months, 12 months | |
| Table 18 | Genetic Abnormalities | Patients with: Any abnormality (n, %) Abnormality in PI3K/Akt/mTOR pathway (n, %) ESR1 abnormality (n, %) | Safety |






REFERENCE SOP: CDS-0102

| Figure<br>No | Description | Variables/Analyses To Be Included | Population |
|---|---|---|---|
| Figure 1 | Overall Survival | Timescale to be used on horizontal axis: ☐ Day ☐ Week ☐ Month ☐ Year | Efficacy Evaluable,<br>Safety |
| Figure 2 | Progression-free Survival | Timescale to be used on horizontal axis: ☐ Day ☐ Week ☐ Month ☐ Year | Efficacy Evaluable,<br>Safety |

| Listing<br>No. | Title | Variables/Analyses To Be<br>Included | Population |
|---|---|---|---|
| 1 | Prior Systemic Therapy | Patient Number Start Date End Date Medication Taken Regimen Number Disease Setting Best Overall Response Reason Therapy Ended - Specify | Enrolled Patients |
| 2 | Current Hormonal Therapy | Patient Number Visit Name Disease Setting Medication Taken Start Date End Date Reason for Therapy End | Enrolled Patients |
| 3 | Biodesix Information | Patient Number Age Sex Race Ethnicity Performance Status at Screening (ECOG) ER (most recent) PR HER 2 Current Endocrine Therapies Prior Endocrine Therapies Prior Adjuvant Therapies Prior Metastatic Therapies Prior Neoadjuvant Therapies Disease Stage at Diagnosis Date of Treatment Start Best Overall Response Date of Best Overall Response PFS (months) OS (months) | Enrolled Patients |
| 4 | Patients with ESR1 Mutation | Patient Number | Safety,<br>whose Tissue Samples<br>were Assessed |
